CLINICAL TRIAL: NCT00072111
Title: Phase I Study of Anakinra Mediated Tumor Regression and Angiogenesis Inhibition in Subjects With Cancers Producing Interleukin-1
Brief Title: Anakinra in Treating Patients With Metastatic Cancer Expressing the Interleukin-1 Gene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000335469; NCI-03-C-0281; NCT00068016 (obsolete NCT alias)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2006-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Biological: anakinra

SUMMARY:
RATIONALE: Biological therapies, such as anakinra, may interfere with the growth of the tumor cells and slow the growth of metastatic tumors that express the interleukin-1 gene.

PURPOSE: This phase I trial is studying the side effects and best dose of anakinra in treating patients with metastatic cancer that expresses the interleukin-1 gene.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of anakinra in patients with metastatic cancer expressing the interleukin-1 gene.
* Determine the steady state pharmacokinetics of this drug in these patients.

Secondary

* Determine the antitumor efficacy of this drug in these patients.
* Determine gene expression changes in tumor biopsies and circulating leukocyte and cytokine levels in these patients before and after treatment with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive anakinra subcutaneously 1-3 times daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of anakinra until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 6 patients are treated at that dose.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic cancer
* Measurable disease

  * Able to be percutaneously biopsied with minimum morbidity on protocol NCI-99-C-0128
* Tumor expression of interleukin-1 by biopsy
* Progressive disease during prior standard first-line chemotherapy OR refused standard first-line chemotherapy
* No active intracranial or leptomeningeal metastases

  * Prior radiotherapy to or resection of intracranial metastatic disease allowed provided there is no evidence of active disease on MRI or CT scan for the past month AND there is no requirement for concurrent anticonvulsant or steroid medications

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 4 months

Hematopoietic

* Platelet count greater than 75,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3

Hepatic

* PT within 2 seconds of the upper limit of normal
* Bilirubin less than 1.5 mg/dL

Renal

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance greater than 30 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* No allergy to proteins made from bacteria
* No active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 30 days since prior biologic therapy
* No concurrent systemic immune modulators

Chemotherapy

* See Disease Characteristics
* More than 30 days since prior chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent steroids

Radiotherapy

* See Disease Characteristics
* More than 14 days since prior localized radiotherapy to non-target lesions and recovered
* More than 30 days since other prior radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 30 days since prior antibiotic therapy for infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Principal Investigator — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States